CLINICAL TRIAL: NCT03748238
Title: Systematic And Standardized Hysteroscopic Endometrial Injury For Treatment Of Recurrent Implantation Failure
Brief Title: Endometrial Injury In Recurrent Implantation Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gurgan Clinic (Network)
Responsible Party: Principal Investigator, Muberra Namlı Kalem, Assoc Professor, MD, Gurgan Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201871
Record Dates: First submitted 2018-11-14; First posted 2018-11-20 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Infertility; Endometrial Diseases
Keywords: Recurrent implantation failure; Endometrial injury; Implantation; Hysteroscopy
MeSH Terms: conditions — Infertility; Uterine Diseases | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injury group (Experimental): Endometrial injury with hysteroscopy
  Interventions: Procedure: Endometrial Injury with Hysteroscopy
- Control group (No Intervention): No hysteroscopy

INTERVENTIONS:
Procedure: Endometrial Injury with Hysteroscopy — All office hysteroscopy procedures will be done transvaginally under sedation with a 5 mm 30 degree lens supplied with a 5 F working channel continuous flow office hysteroscope (Bettocchi office hysteroscope, Karl Storz, Tuttlingen, Germany) without speculum or tenaculum. Briefly, following cervical passage and initial endometrial cavity investigation endometrial injury will be performed without energy modality (i.e. with scissors). Endometrial injury will perform first on the fundus by cutting into the endometrium (without injuring the myometrium) transversally. Later, vertical incisions will perform 0,5 cm apart each other, on the anterior and posterior walls of the uterus, 1-1.5 cm away from the fundus and one cut for each lateral wall
  Arms: Injury group

SUMMARY:
The aim of this study is to investigate that the efficacy of the endometrial injury before IVF in recurrent implantation failure patients.

DETAILED DESCRIPTION:
This is a prospective and randomized controlled trial investigating the effect of hysteroscopic endometrial injury for treatment of recurrent implantation failure. Approximately 230 patients who had failed to achieve a clinical pregnancy after the transfer of at least four good-quality embryos in a minimum of three fresh or frozen cycles to a woman under the age of 40 years will be randomized into two groups. Injury group will receive endometrial injury during their hysteroscopic procedure, whereas the control group (n=115) did not. This study will investigate that, whether the endometrial injury is beneficial in recurrent implantation failure patients to increase the odds of clinical pregnancy rates, live birth rates, and implantation rates.

ELIGIBILITY:
Inclusion Criteria:

* Women under the age of 40 who met the RIF definition
* Patients whose follicle-stimulating hormone (FSH) levels were ≤ 15 IU/mL

Exclusion Criteria:

* Patients with congenital uterine anomalies
* Patients with Asherman's syndrome
* Patients with uterine cavity distorted by myoma or endometrial polyps
* Patients with confirmed endometriosis or endometrioma
* Patients with BMI of <18.5 and >29.9

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women with recurrent implantation failure
Enrollment: 230 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Positive Pregnancy | 1month
  Blood concentration of beta-hcg

CONTACTS AND LOCATIONS:
Overall Officials: Ziya Kalem, MD, Principal Investigator — Gurgan Clinic IVF and Women Health Center; Halil Ruso, Embryologist, Principal Investigator — GurganClinic IVF and Women Health Center; Antonis Makrigiannakis, MD,Professor, Principal Investigator — Greek University
Locations (1):
- Gurgan Clinic IVF and Women Health Center, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No